CLINICAL TRIAL: NCT04694560
Title: A Phase 2 Time-Limited Approach to Front-Line Ibrutinib for Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma Patients Who Achieve Complete Remission or Partial Remission With Undetectable Minimal Residual Disease
Brief Title: A Time-Limited Approach to Treatment With Ibrutinib for Chronic Lymphocytic Leukemia and Small Lymphocytic Lymphoma
Status: Withdrawn | Type: Observational
Why Stopped: Lack of potential participants given the other treatment options currently available to people
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Pharmacyclics LLC. (Industry)
Responsible Party: Sponsor
Other Study IDs: 20-284
Record Dates: First submitted 2020-12-28; First posted 2021-01-05 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2023-03

CONDITIONS: CLL; SLL; CLL/SLL; Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: Small Lymphocytic Lymphoma; Chronic Lymphocytic Leukemia; CLL/SLL; SLL; CLL; Ibrutinib; Ibrutinib monotherapy; anti-CD20 monoclonal antibody; MRD; U-MRD; 20-284; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- CLL/SLL: Diagnosis of CLL or SLL confirmed by the enrolling institution
  Interventions: Other: Treatment Free Observation

INTERVENTIONS:
Other: Treatment Free Observation — Participants without evidence of clinical relapse will remain off therapy and continue serial monitoring through end of study at 24 cycles. Participants with clinical relapse will continue to be monitored off therapy through 24 cycles or until meeting criteria for treatment per iwCLL criteria. If participants experience clinical relapse requiring treatment, radiology assessment, disease assessment, and testing for resistance mutations will be performed. Participants will be observed for an additional 12 cycles following start of reintroduction of therapy.

SUMMARY:
The purpose of this study is to find out whether people with CLL or SLL who are currently receiving treatment with ibrutinib can stop treatment and remain off-treatment for at least 12 months, if they have achieved complete or partial remission of their disease.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18-years-old
* Diagnosis of CLL or SLL confirmed by the enrolling institution
* Negative del(17p) test confirmed by FISH testing prior to initiating treatment with ibrutinib
* Receiving commercial treatment with an ibrutinib-based regimen in the front-line setting as defined below with the intent to discontinue therapy on C1D1:

  1. Ibrutinib monotherapy
  2. Ibrutinib in combination with anti-CD20 monoclonal antibody (Patients must have completed the anti-CD20 monoclonal antibody portion of the regimen prior to signing consent)
* Patients must have received ibrutinib-based therapy for at least 15 months. Dose interruptions and reductions during this treatment period may have been carried out per treating provider discretion.
* Response evaluation performed by radiology assessment (CT or MRI imaging of neck / chest / abdomen / pelvis) confirming complete remission or partial remission by iwCLL criteria.
* Peripheral blood (by flow cytometry per institutional standards) testing for MRD confirming U-MRD to a sensitivity of 10^-4. MRD testing must be confirmed to follow ERIC consensus criteria.

  1. CR with or without U-MRD in peripheral blood
  2. PR with U-MRD in peripheral blood

Exclusion Criteria:

* Any life-threatening illness, medical condition, or organ system dysfunction that, in the investigator's opinion, could compromise the subject's safety or put the study outcomes at undue risk..
* Unwilling or unable to participate in all required study evaluations and procedures. Unable to understand the purpose and risks of the study and to provide a signed and dated informed consent form (ICF) and authorization to use protected health information (in accordance with national and local patient privacy regulations).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Potential research subjects will be identified by a member of the patient's treatment team, the protocol investigator, or research team at Memorial Sloan-Kettering Cancer Center (MSKCC). If the investigator is a member of the treatment team, s/he will screen their patient's medical records for suitable research study participants and discuss the study and their potential for enrolling in the research study. Potential subjects contacted by their treating physician will be referred to the investigator/research staff of the study. The principal investigator may also screen the medical records of patients with whom they do not have a treatment relationship for the limited purpose of identifying patients who would be eligible to enroll in the study and to record appropriate contact information in order to approach these patients regarding the possibility of enrolling in the study.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-12-22 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-03-06 (Actual)

PRIMARY OUTCOMES:
Tumor Free Survival rate | At the end of Cycle 24 (each cycle is 28 days) cycles +/- 14 days
  Participants will be evaluated by iwCLL / International Workshop on Chronic Lymphocytic Leukemia criteria

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Mato, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (2):
- United States (2):
  - Atrium Health (Data Collection Only), Monroe, North Carolina
  - University of Pennsylvania (Data Collection Only), Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org